CLINICAL TRIAL: NCT05191459
Title: Are There Any Differences in Occurrence of Lung Changes Associated With the Chronic Heart Failure Between the Patients With Preserved and Reduced Ejection Fraction of Left Ventricle?
Brief Title: Impact of Hear Failure on Lungs in Patients With Heart Failure
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Marta Dąbrowska, Principal Investigator, Medical University of Warsaw
Other Study IDs: Lungs in heart failure
Record Dates: First submitted 2022-01-02; First posted 2022-01-13 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure
Keywords: heart failure; lung function; chest computed tomography
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Heart failure and preserved ejection fraction: 42 patients 50-90 years with preserved ejection fraction (EF ≥50%)
- Heart failure and reduced ejection fraction: 42 patients 50-90 years with reduced ejection fraction ((EF≤40%)

SUMMARY:
Heart failure (HF) is a common disease, which impacts on other organs. Despite an ongoing progress in knowledge about HF, there are still some uncharted aspects of impact of HF on respiratory system. The aim of the study is to determine whether there are any differences in pulmonary changes assessed in chest CT, chest ultrasound or in pulmonary function tests between patients with HF with decreased (≤40%; HFrEF) and preserved (≥50%; HFpEF) ejection fraction.

Eighty four patients diagnosed with HF will be included (42 with HFrEF and 42 with HFpEF) and the following tests will be performed :

1. echocardiography
2. chest X-ray and CT
3. assessment of lung hydration in ultrasound
4. spirometry, plethysmography, diffusion capacity for carbon monoxide (DLCO)
5. arterial blood gas analysis
6. peripheral blood collection

In patients with abnormal, suspected changes in the lungs diagnosed in the chest CT bronchoscopy and endobronchial ultrasound (EBUS) will be offered.

The primary outcome will be difference in frequency of chest CT abnormalities (ground-glass opacities or interlobular septal thickening or pleural effusion or mediastinal lymphadenopathy) between patients with HFrEF and HFpEF

The secondary outcomes will be:

1. difference in pulmonary function test results (FEV1, FVC, TLC, RV, DLCO)
2. differences in arterial pO2 and pCO2
3. differences in B- line scores in ultrasound
4. differences in concentration of blood biomarkers (troponin, CRP, NTproBNP, IL-6, TNF-α, sST2, Gal-3, GDF-15)

The results of the study will allow to .better understand the pathomechanisms of the occurrence of lesions in lungs secondary to HF. Thus, it may anable to reduce unnecessary diagnostics in patients with HF in the future.

DETAILED DESCRIPTION:
Heart failure (HF) is a global disease, which affects 1-2% adults worldwide. It is believed that 60% of these patients have HF with reduced ejection fraction (EF≤40%; HFrEF), 24% have HF with mildly reduced (EF 41-49%; HFmrEF) and 16% have HF with preserved ejection fraction (EF ≥50%, HFpEF). Despite its high prevalence, there are still many aspects of the disease that are not well recognized yet. One of them is impact of HFpEF on function lungs. Previous studies focused on this topic are scarce and mainly concern patients with advanced HFrEF. It was documented that HFrEF may lead to both lung abnormal changes in chest imaging and lung function tests. It may sometimes lead to unnecessary diagnostic procedures. However, pathophysiology and clinical relevance between heart and lung function in HFpEF patients still need to be elucidated.

Thus the aim of the study is to determine whether pulmonary abnormal findings found both in chest imaging and pulmonary function tests are comparable in patients with HFpEF and HFrEF.

Patients:

The study will include 84 patients (42 with HFrEF and 42 with HFpEF) aged 50-90 years diagnosed with chronic HF (NYHA II/III) in a stable period.

Inclusion criteria:

1. Age: 50-90 years old
2. Chronic heart failure (NYHA class II-III)
3. Signed informed consent

Exclusion Criteria:

1. No consent to the study
2. Age: <50 or >90 years old
3. Any chronic pulmonary diseases diagnosed before
4. Acute respiratory infection 14 days before enrollment (fever ≥38°C and at least one additional symptoms of infection)
5. Acute kidney injury or chronic kidney failure (stage 4 or 5)
6. Acute hepatic failure

Power analysis and sample size calculations indicated that a sample size of 84 subjects would provide 80% statistical power to detect significant differences between the two groups (alpha = 0.05, beta = 0.20) assuming that abnormal findings in chest CT will be present in 60% of patients with HFrEF and in 30% of subjects with HFpEF.

Included patients will be examined by:

1. echocardiographic examination of the heart
2. X-ray and CT of the chest
3. spirometry, plethysmography, diffusion capacity for carbon monoxide (DLCO)
4. arterial blood gas testing
5. assessment of lung hydration in ultrasound
6. peripheral blood collection In patients with abnormal, suspected changes in the lungs revealed in the chest CT bronchoscopy and endobronchial ultrasound (EBUS) will be considered.

The primary outcome :

1. difference in frequency of chest CT abnormalities (ground-glass opacities or interlobular septal thickening or pleural effusion or mediastinal lymphadenopathy) between patients with HFrEF and HFpEF

The secondary outcomes:

1. difference in pulmonary function test results (FEV1, FVC, TLC, RV, DLCO)
2. differences in arterial pO2 and pCO2
3. differences in B- line score in lung ultrasound
4. differences in concentration of blood biomarkers (troponin, CRP, NTproBNP, IL-6, TNF-α, sST2, Gal-3, GDF-15)

The results of the study will allow to better understand the pathomechanisms of the occurrence of lesions in lungs secondary to HF. Thus, it may enable to reduce unnecessary diagnostics in patients with HF in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 50-90 years old
2. Chronic heart failure (NYHA class II-III)
3. Signed informed consent

Exclusion Criteria:

1. No consent to the study
2. Age: <50 or >90 years old
3. Any chronic pulmonary diseases diagnosed before
4. Acute respiratory infection 14 days before enrollment (fever ≥38°C and at least one additional symptoms of infection)
5. Acute kidney injury or chronic kidney failure (stage 4 or 5)
6. Acute hepatic failure

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic heart failure between 50-90 years old.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
difference in frequency of chest CT abnormalities between patients with HFrEF and HFpEF | baseline
  difference in frequency of chest CT abnormalities (ground-glass opacities or interlobular septal thickening or pleural effusion or mediastinal lymphadenopathy) between patients with HFrEF and HFpEF

SECONDARY OUTCOMES:
Differences in lung function measured in spirometry between patients with HFpEF and HFrEF | baseline
  Differences in median forced expiratory volume in 1st second (FEV1) and forced volume capacity (FVC) in spirometry between patients with HFpEF and HFrEF
Differences in lung function measured by bodypletysmography between patients with HFpEF and HFrEF | baseline
  Differences in median total lung capacity (TLC) and reserved volume(RV) in body plethysmography between patients with HFpEF and HFrEF
Difference in DLCO between patients with HFpEF and HFrEF | baseline
  Differences in median diffusing capacity of the lungs for carbon monoxide (DLCO) between patients with HFpEF and HFrEF
Differences in arterial pO2 and pCO2 between patients with HFpEF and HFrEF | baseline
  Differences in median arterial pO2 and pCO2 between patients with HFpEF and HFrEF
Differences in lung hydration between patients with HFpEF and HFrEF | baseline
  difference in median B- line score in lung ultrasound between patients with HFpEF and HFrEF

CONTACTS AND LOCATIONS:
Overall Officials: Marta Dąbrowska, Principal Investigator — Medical University of Warsaw
Locations (1):
- Department of Internal Medicine, Pulmonary Diseases and Allergy, Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cardinale L, Priola AM, Moretti F, Volpicelli G. Effectiveness of chest radiography, lung ultrasound and thoracic computed tomography in the diagnosis of congestive heart failure. World J Radiol. 2014 Jun 28;6(6):230-7. doi: 10.4329/wjr.v6.i6.230. PMID 24976926
- [Background] Kee K, Naughton MT. Heart failure and the lung. Circ J. 2010 Nov;74(12):2507-16. doi: 10.1253/circj.cj-10-0869. Epub 2010 Oct 28. PMID 21041971
- [Background] Ardekani MS, Issa M, Green L. Diagnostic and economic impact of heart failure induced mediastinal lymphadenopathy. Int J Cardiol. 2006 Apr 28;109(1):137-8. doi: 10.1016/j.ijcard.2005.04.011. No abstract available. PMID 16574532
- [Background] Obokata M, Olson TP, Reddy YNV, Melenovsky V, Kane GC, Borlaug BA. Haemodynamics, dyspnoea, and pulmonary reserve in heart failure with preserved ejection fraction. Eur Heart J. 2018 Aug 7;39(30):2810-2821. doi: 10.1093/eurheartj/ehy268. PMID 29788047
- [Background] Huang WM, Feng JY, Cheng HM, Chen SZ, Huang CJ, Guo CY, Yu WC, Chen CH, Sung SH. The role of pulmonary function in patients with heart failure and preserved ejection fraction: Looking beyond chronic obstructive pulmonary disease. PLoS One. 2020 Jul 7;15(7):e0235152. doi: 10.1371/journal.pone.0235152. eCollection 2020. PMID 32634145
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992